CLINICAL TRIAL: NCT00672178
Title: Phase I/II Trial Evaluating Toxicity and Efficacy of Adding Stereotactic Body Radiotherapy to Sorafenib in Patients With Metastatic, Recurrent, or Unresectable Renal Cell Cancer
Brief Title: Stereotactic Body Radiotherapy (SBRT) and Sorafenib in Patients With Metastatic, Recurrent, or Unresectable Renal Cell Cancer (RCC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Duke University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001398
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Renal Cell Carcinoma
Keywords: RCC; metastatic; sorafenib
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Stereotactic body radiation — Stereotactic body radiotherapy will be given in three cohorts of increasingly higher dose levels: Cohort 1: 6 Gy/fraction x 3 fractions (total=18 Gy) over 5 days; Cohort 2: 8 Gy/fraction x 3 fractions over 5 days; Cohort 3: 10 Gy/fraction x 3 fractions over 5 days.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of combined stereotactic body radiotherapy (SBRT) + sorafenib in the treatment of patients with Stage IV renal cell carcinoma (RCC) who have recurred locally, developed progression of an unresectable primary or progression of extra-cranial and/or extra-pulmonary metastases while on sorafenib. All subjects will remain on sorafenib during SBRT.

DETAILED DESCRIPTION:
In the phase I portion of this investigation, subjects will be enrolled in cohorts of three to the SBRT dose groups. Subjects will remain on sorafenib therapy during SBRT. Any change in sorafenib dosage before, during or after SBRT will be at the discretion of the subject's medical oncologist. Subjects will be assessed during, immediately after and at 4 and 8 weeks post-therapy for toxicity.

Stereotactic body radiotherapy will be given in increasingly higher dose levels each cohort until the maximum tolerated dose of radiation is determined.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Zubrod Performance Status 0 or 1
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin > 9.0 g/dl
  * Absolute neutrophil count (ANC) > 1,500/mm3
  * Platelet count > 100,000/mm3
  * Total bilirubin < 1.5 times institutional upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 times the institutional ULN
  * Creatinine < 1.5 times institutional ULN
* Histologically or cytologically confirmed renal cell carcinoma, which is metastatic, unresectable or recurrent.
* Life expectancy > 6 months
* Local recurrence or progression of primary lesion or progression, or symptomatic progression in extra-cranial, extra-pulmonary metastases while on sorafenib
* Measurable disease
* Bone metastases must have a tissue component measurable by imaging.
* No untreated brain metastases
* Resolution of pre-existing toxicity from prior therapy excluding alopecia and taste alteration.
* Willingness and ability to comply with continuing sorafenib, visits, treatment plans, laboratory tests and study procedures.
* All treated lesions must comply with SBRT dose constraints
* More than 28 days since any prior systemic or local therapy for this cancer, including investigational agents and surgical procedures exclusive of sorafenib
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control)
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Ability to understand and the willingness to sign a written informed consent.
* Prothrombin time(PT) and partial thromboplastin time (PTT) within normal limits.

Exclusion Criteria:

* Lesion in remaining (solo) kidney
* Contraindications to radiotherapy or prior radiotherapy overlapping current site(s) of disease.
* Cardiac disease: Congestive heart failure. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding problems
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkpatrick, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: Jan 2008-Sept 2009. Study stopped early due to low accrual
Groups:
- SBRT: Stereotactic body radiotherapy concurrent with sorafenib
Period: Overall Study
Arm/Group | SBRT
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SBRT
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Complete and Partial Response (CR+PR)
Time Frame: 8 weeks
Arm/Group | SBRT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | SBRT
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination due to low accrual, only one subject enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No